CLINICAL TRIAL: NCT00411333
Title: Vascular Remodeling and the Effects of Angiogenic Inhibition in Diabetic Retinopathy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R01 EY017528-0; R01EY017528 (NIH)
Record Dates: First submitted 2006-12-13; First posted 2006-12-14 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-11

CONDITIONS: Diabetic Retinopathy
Keywords: diabetic retinopathy; fluorescein angiography; steroid; anti-angiogenesis
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Triamcinolone Acetonide

INTERVENTIONS:
Drug: triamcinolone acetonide (Kenalog)

SUMMARY:
The retinal vasculature changes dramatically in patients with diabetic retinopathy especially between non-proliferative and proliferative disease. The retinal vasculature can be imaged and quantified using special dyes. This study will test whether the pattern of the retinal vasculature changes in patients with different levels of diabetic retinopathy can be quantified using computerized image analysis. In addition, the study will evaluate whether new drugs to treat diabetic retinopathy will be able to reverse these vascular changes.

DETAILED DESCRIPTION:
In this study, we are studying whether vascular density decreases during diabetic retinopathy prior to the pathological neovascularization seen in proliferative disease that results in blindness in more than 50 percent of patients, and whether the adverse, early vascular remodeling and neovascularization can be reversed by anti-angiogenic therapeutics. We have shown that vascular density decreases during early stages of diabetic retinopathy, prior to the pathological neovascularization that defines proliferative retinopathy, and that this change may be reversible with new anti-angiogenic therapeutics. To test this hypothesis we will determine (1) how blood vessels remodel and whether vascular density truly decreases during diabetic retinopathy and (2) how the anti-angiogenic steroid triamcinolone acetonide affects vascular density and pattern during human diabetic retinopathy and in our experimental model, the avian CAM model.

Twenty patients (n = 20) for each of the 4 NPDR stages will be enrolled. In addition, a control group of 20 normal subjects will be recruited from the same clinical practice that do not have diabetes and no evidence of any vascular disease, for a total of 100 patients in the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

- Presence of mild, moderate, severe, or very severe non-proliferative diabetic retinopathy (defined as ETDRS level >10) in at least one eye (based on ETDRS criteria)

Exclusion Criteria:

* Any condition that might impair the patient's ability to give informed consent
* Any condition or media opacity that might impair the patient's ability to perform vision tests, color fundus photographs or fluorescein angiography
* Severe allergy or other contraindication to sodium fluorescein dye
* Participating in any other ophthalmic clinical trial

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Change in retinal vascular density from baseline on fluorescein angiography

SECONDARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Peter K Kaiser, MD, Principal Investigator — Cole Eye Institute
Locations (1):
- Cole Eye Institute, Cleveland, Ohio, United States

REFERENCES:
- [Result] Parsons-Wingerter P, Radhakrishnan K, Vickerman MB, Kaiser PK. Oscillation of angiogenesis with vascular dropout in diabetic retinopathy by VESsel GENeration analysis (VESGEN). Invest Ophthalmol Vis Sci. 2010 Jan;51(1):498-507. doi: 10.1167/iovs.09-3968. Epub 2009 Sep 24. PMID 19797226
- [Result] Vickerman MB, Keith PA, McKay TL, Gedeon DJ, Watanabe M, Montano M, Karunamuni G, Kaiser PK, Sears JE, Ebrahem Q, Ribita D, Hylton AG, Parsons-Wingerter P. VESGEN 2D: automated, user-interactive software for quantification and mapping of angiogenic and lymphangiogenic trees and networks. Anat Rec (Hoboken). 2009 Mar;292(3):320-32. doi: 10.1002/ar.20862. PMID 19248164